CLINICAL TRIAL: NCT01057108
Title: A Double Blind, Randomized, Placebo Controlled Trial to Evaluate the Efficacy and Safety of FOSTRAP Chewing Gum in Patients With Chronic Kidney Disease and Hyperphosphatemia.
Brief Title: Double Blind Randomized Placebo Controlled Trial of FOSTRAP Chewing Gum in Patients With CKD and Hyperphosphatemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Denver Nephrologists, P.C. (Other)
Collaborators: CM&D Pharma Limited (Industry)
Responsible Party: Geoffrey A. Block, MD/ Principal Investigator, Denver Nephrologists, PC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMD 002
Record Dates: First submitted 2010-01-25; First posted 2010-01-27 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2011-01

CONDITIONS: Hyperphosphatemia; Chronic Kidney Disease
Keywords: Hyperphosphatemia; chronic kidney disease; salivary phosphorus
MeSH Terms: conditions — Hyperphosphatemia; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ESRD: FOSTRAP Chewing Gum (Active Comparator)
  Interventions: Other: FOSTRAP Chewing Gum
- CKD: FOSTRAP Chewing Gum (Active Comparator)
  Interventions: Other: FOSTRAP Chewing Gum
- ESRD Matching Placebo (Placebo Comparator)
  Interventions: Other: Placebo chewing gum
- CKD Matching Placebo (Placebo Comparator)
  Interventions: Other: Placebo chewing gum

INTERVENTIONS:
Other: FOSTRAP Chewing Gum — 20 mg BID
  Arms: ESRD: FOSTRAP Chewing Gum
Other: FOSTRAP Chewing Gum — 40 mg BID
  Arms: ESRD: FOSTRAP Chewing Gum
Other: FOSTRAP Chewing Gum — 20 mg TID
  Arms: CKD: FOSTRAP Chewing Gum
Other: FOSTRAP Chewing Gum — 20 mg TID
  Arms: ESRD: FOSTRAP Chewing Gum
Other: Placebo chewing gum
  Arms: CKD Matching Placebo; ESRD Matching Placebo

SUMMARY:
The phosphorus content in saliva is increased in chronic kidney disease. We hypothesize that a chewing gum that binds salivary phosphorus would be a novel, effective agent to reduce serum levels of phosphorus in patients with chronic kidney disease. We are testing this hypothesis using a chewing gum called FOSTRAP which has been shown to be effective in a small, non-randomized study in patients with chronic kidney disease on hemodialysis.

DETAILED DESCRIPTION:
A double-blind, randomized, placebo, controlled trial with an open label extension for those subjects with end stage renal disease (ESRD).

Patients with ESRD will be randomized to receive either FOSTRAP™ 20 mg BID, FOSTRAP™ 40 mg BID or matching placebo 2x/day. All subjects will participate in a 4 week chewing period followed by a 4 week follow up period. All subjects will then enter an open label 2 week extension phase in which they will receive FOSTRAP™ 20 mg TID.

Patients with chronic kidney disease (CKD) not on dialysis will receive either FOSTRAP™ 20 mg 3x/day or placebo TID for 4 weeks followed by a 4 week follow up period.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women > 18 years of age;
2. The subject has voluntarily signed and dated the most recent informed consent form approved by an Institutional Review Board (IRB);
3. The subject will, in the opinion of the investigator, be compliant with prescribed therapy;
4. Subject must be able to communicate and be able to understand and comply with the requirements of the study;
5. For subjects with CKD not on dialysis- kidney function at any stage that in the opinion of the investigator is stable and not expected to initiate dialysis within 3 months;
6. For subjects with CKD not on dialysis- a screening serum phosphorus value greater than or equal to 4.5 mg/dL;
7. For subjects with ESRD - a screening serum phosphorus value greater than or equal to 4.6 mg/dL and less than or equal to 9.0 mg/dL and one of the two conditions: A mean historical value of the most recent 2 phosphorus measurements ≥ 4.6 and less than or equal to 9.0 mg/dL at the time of written informed consent or A second screening serum phosphorus value greater than or equal to 4.6 mg/dL and less than or equal to 9.0 mg/dL performed not less than 7 days from the date of the previous screening;
8. In the opinion of the investigator, subjects with ESRD must be prescribed a stable dialysis regimen (3x/week) for ≥ 4 weeks prior to baseline and must have a stable dialysis access;
9. Subjects with ESRD must have an historical URR ≥ 65% for at least 4 weeks prior to baseline;
10. All subjects must have NO change in prescribed dose or frequency of any of the following medications ≥ 14 days prior to baseline:

    1. Phosphate binding products including prescribed and over-the counter
    2. Oral or injectable active vitamin D
    3. Oral nutritional vitamin D
    4. Calcimimetics
    5. Calcium supplements
    6. Anti-osteoporotic medication (e.g. bisphosphonates)
11. Subject must be prescribed a diet appropriate for patients with their stage of kidney disease, and must be willing to avoid intentional changes in diet; and
12. Subjects must have a screening salivary flow rate by Saxon test ≥ 1 g/2 min.

Exclusion criteria:

1. Receiving or has received an investigational product (or is currently using an investigational device) within 28 days prior to baseline;
2. Known sensitivity to chitin or allergy to shellfish;
3. Clinical evidence of active malignancy and/or receiving systemic chemotherapy/radiotherapy with the exception of basal cell or squamous carcinoma of the skin;
4. Clinically significant infection requiring treatment with antibiotics (within 7 days prior to baseline);
5. Inpatient hospitalization within 14 days prior to baseline with the exception of hospitalizations related to vascular access procedures;
6. Planned surgical intervention for secondary hyperparathyroidism;
7. In the opinion of the investigator, inability to chew gum for 60 minutes;
8. Planned relocation to another area within the next 4 months;
9. Subject has a known history of immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result;
10. Active drug or alcohol dependence or abuse (excluding tobacco use) in the opinion of the principal investigator;
11. Unstable medical condition which in the opinion of the investigator would compromise successful completion of the study;
12. Known active liver disease with AST or ALT levels greater than 3X the upper limit of normal; and
13. Subject has had a major cardiovascular event within 90 days of screening. The investigator should be guided by evidence of any of the following;

    1. Acute myocardial infarction
    2. Acute cerebral vascular event
    3. Vascular surgical intervention
    4. Coronary Revascularization
    5. Decompensated congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Change in serum phosphorus from baseline to Day 29 | Day 1 and Day 29

SECONDARY OUTCOMES:
Change in salivary phosphorus from baseline to Day 29 | Day and Day 29
Proportion of subjects whose serum phosphorus reduction from baseline to Day 29 is greater than or equal to 0.5 mg/dL | Day 1 and Day 29
Proportion of subjects whose serum phosphorus reduction from baseline to Day 29 is greater than or equal to 1.5 mg/dL | Day 1 and Day 29
Change in serum phosphorus from Day 57 to day 71 for subjects with ESRD | Day 57 and Day 71
For subjects with ESRD absolute and relative difference between serum phosphorus (baseline to Day 29)- (Day 57 to day 71) | Day 29, Day 57, Day 71
Change in salivary phosphorus from Day 57 to Day 71 | Day 57 and Day 71

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey A Block, MD, Principal Investigator — Denver Nephrologists, PC
Locations (1):
- Denver Nephrologists, PC, Denver, Colorado, United States

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Block GA, Persky MS, Shamblin BM, Baltazar MF, Singh B, Sharma A, Pergola P, Smits G, Comelli MC. Effect of salivary phosphate-binding chewing gum on serum phosphate in chronic kidney disease. Nephron Clin Pract. 2013;123(1-2):93-101. doi: 10.1159/000351850. Epub 2013 Jun 22. PMID 23797006